CLINICAL TRIAL: NCT01543386
Title: Effects of Curcumin Loading Dose on Vascular Reactivity of Healthy Middle-aged Smokers
Brief Title: Effects of Curcumin on Vascular Reactivity
Acronym: CURCUMIN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Association Régionale de Cardiologie d'Auvergne (Unknown); ARDEC Association de Recherche de Développement et d'Enseignement de la Cardiologie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0113
Record Dates: First submitted 2012-02-16; First posted 2012-03-05 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers (Middle-aged Smokers)
Keywords: Polyphenol; Curcumin; Endothelium, vascular; Endothelium-dependant relaxing factor; Smoking; Transcriptome
MeSH Terms: conditions — Smoking | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- curcumin (Other): The aim of this study is to determine if an oral loading-dose of curcumin can improve vascular endothelium reactivity in patients with moderate cardiovascular risk
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin — The aim of this study is to determine if an oral loading-dose of curcumin can improve vascular endothelium reactivity in patients with moderate cardiovascular risk

SUMMARY:
The aim of this study is to determine if an oral loading-dose of curcumin can improve vascular endothelium reactivity in patients with moderate cardiovascular risk

DETAILED DESCRIPTION:
The aim of this study is to determine if an oral loading-dose of curcumin can improve vascular endothelium reactivity in patients with moderate cardiovascular risk

ELIGIBILITY:
Inclusion Criteria:

* 50 to 70 year-old volunteers
* smokers

Exclusion Criteria:

* treated hypertension
* treated hypercholesterolemia
* chronic disease
* vegetarian or other unusual diets
* chronic alcoholism

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Changes in brachial Flow Mediated Dilatation | at Visit 1 (Day 0) and visit 2 (Day3/day5)

SECONDARY OUTCOMES:
Changes in fingertip arterial tonometry | at visit 1 (day 0) and visit 2 (day3/day5)
Modifications of leukocytes transcriptome | at visit 1 (day 0) and visit 2 (day3/day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-René LUSSON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Barber-Chamoux N, Milenkovic D, Verny MA, Habauzit V, Pereira B, Lambert C, Richard D, Boby C, Mazur A, Lusson JR, Dubray C, Morand C. Substantial Variability Across Individuals in the Vascular and Nutrigenomic Response to an Acute Intake of Curcumin: A Randomized Controlled Trial. Mol Nutr Food Res. 2018 Mar;62(5). doi: 10.1002/mnfr.201700418. Epub 2018 Feb 12. PMID 29034576